CLINICAL TRIAL: NCT00700453
Title: Video Game-Brain Functioning Reversibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indiana University (Other)
Collaborators: The Center for Successful Parenting Video Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0804-07
Record Dates: First submitted 2008-06-11; First posted 2008-06-18 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-04

CONDITIONS: Brain Functioning and Violent Video Game Play
MeSH Terms: interventions — Control Groups; Cognitive Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control 1 Group (Active Comparator): Subjects randomized to the Control 1 group will abstain from playing any video games for the entire study participation.
  Interventions: Behavioral: Control group with no video game play
- VG1- Control 2 Group (Active Comparator): Subjects randomized to the Control 2 group will play a selected violent video game for 60-120 minutes/day during week 2 of the study and will abstain from any video game play during week 3 of the study.
  Interventions: Behavioral: control 2
- VG1- VG2 group (Active Comparator): Subjects randomized for VG1-VG2 group will play 60-120 minutes/day of a violent video game during weeks 2 & 3 of study participation.
  Interventions: Behavioral: VG1 group (2 weeks of violent video game play)
- VG1-CT group (Active Comparator): Subjects randomized to the VG1-CT group will play 60-120 minutes of a selected violent video game during week 2 of the study and play a selected computerized cognitive training program for 60-120 minutes/day during week 3 of the study.
  Interventions: Behavioral: Cognitive Training

INTERVENTIONS:
Behavioral: Control group with no video game play — Subjects will abstain from all video game play during study participation.
  Other Names: Control 1 group
  Arms: Control 1 Group
Behavioral: control 2 — Subjects will play 1 week of violent video game play followed by 1 week of no video game play.
  Other Names: Control 2 group
  Arms: VG1- Control 2 Group
Behavioral: VG1 group (2 weeks of violent video game play) — Subjects will play a violent video game for 2 weeks of study participation.
  Other Names: VG1-VG2
  Arms: VG1- VG2 group
Behavioral: Cognitive Training — Subjects will play a violent video game for 1 week followed by 1 week of Cognitive Training program.
  Other Names: VG1-CT group
  Arms: VG1-CT group

SUMMARY:
1. Young adults who are exposed to 7-10 days of play of violent video games will show reduced activation in certain regions of the dorsolateral prefrontal cortex and anterior cingulate cortex.
2. Young adults who are exposed to 7-10 days of violent video games will show increased activation in regions of the amygdala.
3. Young adults who abstain from violent video games for a week, after 7-10 days of play of violent video games, will show increased activation of regions in the dorsolateral prefrontal cortex and anterior cingulate cortex and decreased activation of the amygdala, on pre-post fMRI and compared to young adults who continue to play violent video games.
4. Young adults who complete a computerized attention-training program after 7-10 days of violent video games will show increased activation of regions in the dorsolateral prefrontal cortex and anterior cingulate cortex and decreased activation of the amygdala, on pre-post fMRI and compared to young adults who continue to play violent video games.

DETAILED DESCRIPTION:
After an initial screening visit (Visit 1) followed by a one-week period of monitoring their usual media habits, subjects will have a baseline functional magnetic resonance imaging (fMRI) scan (Visit 2). They will then be assigned in a 3:1 ratio to either one-week of violent video game play for 1-2 hours per day or no video game play for one week. Subjects will receive a second fMRI scan at the end of that week (Visit 3). Subjects who had played violent video games will then be assigned to one of three conditions (continued regular violent video game play, no video game play, or an intervention involving cognitive training of working memory) for one week, in order to investigate the persistence of any changes that are found after the first week of exposure. Subjects who had not played video games during the first week will continue to not play video games for the second week. Following that week, subjects will receive a third fMRI scan (Visit 4). One week after the third fMRI scan, subjects will have a final visit or phone call to check on the possibility of any issues with aggressive thoughts/feelings/behavior following the video game exposure in the study (Visit 5). Brain functioning will be measured using functional magnetic resonance imaging (fMRI) as the primary measurement methodology, with neuropsychological testing used as a secondary measurement methodology.

ELIGIBILITY:
Inclusion Criteria:

1. Have K-BIT-2 Matrices IQ>70.
2. Must be 18-29 years old for the entire study.
3. Only males will participate in the study.
4. Must be judged by the investigator to be reliable and cooperative for clinic visits and procedures.
5. Must speak English, be proficient in spoken and written English, and have an educational level and understanding of English required to complete all tests and questionnaires. This is important because some of the tests require automatic and rapid processing of written English.
6. Must have a baseline level of violent video game play averaging less than or equal to 2 hours per week in the year prior to the study, and must have a baseline level of total video game play averaging less than or equal to 5 hours per week in the year prior to the study. These values are based on research by Kronenberger et al. (2005a) showing that nonviolent control adolescent subjects averaged about 2-3 hours of video game play in a week (of which 1-2 hours are spent with violent video games), compared to aggressive adolescent subjects, who averaged about 4-7 hours of video game play per week (of which 3-4 hours are spent with violent video games). Green and Bavalier (2003) based their selection criteria for "action video game players" (VGP) on an average of 1 hour per day for 4 days a week of violent/action video game play and found differences between the VGP group and a non-VGP group on visual processing. It is important to select subjects who are not frequent game players in order for the experimental manipulation (8-16 hours of violent video game play) to be different from their baseline behavioral habits.
7. Must be willing to make lifestyle changes about media habits during the 3-5 week duration of the study.
8. Must have basic level of proficiency with computer to load and play video games.

Exclusion Criteria:

1. Organic brain conditions or seizure disorder (history of febrile seizures with no neurological sequelae is acceptable).
2. Any physical condition or risk that would preclude or invalidate an MRI.
3. Any current mental health diagnosis (other than Adjustment Disorder), based on the Adult Inventory - 4 and follow-up questions from the interviewer, which would be defined as moderate or more severe using the Clinical Global Index - Severity.
4. Treatment of a behavioral or emotional problem (excluding normal adjustment issues, such as adjustment to divorce) by a mental health professional in the past year.
5. Any historical diagnoses of Attention-Deficit/Hyperactivity Disorder, Conduct Disorder, Oppositional-Defiant Disorder, Bipolar Disorder, Schizophrenia (or other disorder involving psychosis), Personality Disorders, or Pervasive Developmental Disorders.
6. Any history of Attention-Deficit/Hyperactivity Disorder, Conduct Disorder, Oppositional-Defiant Disorder, Bipolar Disorder, Schizophrenia (or other disorder involving psychosis), Personality Disorders, or Pervasive Developmental Disorders in first degree relatives (mother, father, siblings, children).
7. Current diagnosis of Substance Abuse or Dependence
8. Use of psychotropic medication for treatment of a mental or behavioral disorder at any time in the study or in the year prior to the study.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-03 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging | Completed at visit 2, 3, and 4 (each visit 7-10 days apart)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent P Mathews, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Radiology-- Research 2 building, Indianapolis, Indiana
  - Riley Outpatient Center Rm 4300, Indianapolis, Indiana

REFERENCES:
- See also: Indiana University; Department of Psychiatry — http://www.iupui.edu/~psych